CLINICAL TRIAL: NCT00176553
Title: A Pilot Study of Dextromethorphan for the Prevention and Treatment of Methotrexate Neurotoxicity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Peter Cole, Cancer Institute of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 3708; CINJ#110113
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Neurotoxicity Syndromes
Keywords: methotrexate neurotoxicity
MeSH Terms: conditions — Neurotoxicity Syndromes | interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dextromethorphan — Patients will receive an inert carrier with or without dextromethorphan. The study drug will be administered at 1.5 mg/kg/dose on a BID schedule. The first dose to be given prior to each scheduled intravenous and/or intrathecal administration of methotrexate and continued for a total of seven days.

SUMMARY:
The purposes of this study are to find out whether dextromethorphan can prevent the short or long-term neurologic side effects of methotrexate, and whether dextromethorphan can improve symptoms of short-term neurologic side effects if they do occur.

DETAILED DESCRIPTION:
We believe that we are beginning to understand the biological cause of the neurotoxicity that happens after treatment with methotrexate. Dextromethorphan, an ingredient in common cough medicines, may be able to prevent and/or treat this neurotoxicity. We have given dextromethorphan to a small group of patients who developed severe neurologic side effects after methotrexate. All had a complete recovery within one day.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed acute lymphocytic leukemia (ALL), non-Hodgkin's lymphoma (NHL) or OS. Patients will be separately stratified and randomized by disease.
* Patients with history of seizures are eligible but will be stratified separately.

Exclusion Criteria:

* Patients taking monoamine oxidase inhibitors (MAOIs) will be excluded from the study, because of the risk of severe drug interactions.
* Pregnant or lactating women.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2003-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To determine whether dextromethorphan decreases the subacute toxicities associated with intravenous and intrathecal methotrexate | 5 years

SECONDARY OUTCOMES:
To determine whether dextromethorphan can alleviate acute or subacute neurotoxicity when it does occur after intravenous or intrathecal methotrexate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Cole, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Cancer Institute of New Jersey, New Brunswick, New Jersey, United States